CLINICAL TRIAL: NCT05154903
Title: Citicoline in Acute Ischemic Stroke
Brief Title: Citicoline in Ischemic Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hossam Shokri, prof, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5555
Record Dates: First submitted 2021-10-06; First posted 2021-12-13 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Acute Ischemic Stroke
Keywords: citicoline; Egypt; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Intervention Model Description: This is a Prospective Randomized Open label trial with Blinded Evaluators, Citicoline will be administered in continuous iv infusion in a dose of 2000 mg per day for the first week following AIS then by oral route for the next 5 weeks.
  The number of patients needed for this proposal is 200 (100 per group): group 1 (citicoline) : receiving citicoline and group 2 (control) not receiving citicoline. A 10% increase will be expected to avoid possible drop-outs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citicoline (Active Comparator): the Citicoline group will receive citicoline in continuous Iv infusion in a dose of 2000 mg per day for the first week following AIS then by oral route for the next 5 weeks
  Interventions: Drug: Citicoline 500 MG
- control (No Intervention): the control group will not receive citicoline

INTERVENTIONS:
Drug: Citicoline 500 MG — Citicoline will be administered in continuous iv infusion in a dose of 2000 mg per day for the first week following AIS then by oral route for the next 5 weeks.
  Arms: Citicoline

SUMMARY:
There is evidence that citicoline is the only neuroprotectant able to improve the functional status of the patients after an acute ischemic stroke.

Citicoline is a neuroprotectant drug against cerebral ischemia, with positive results, both in experimental and clinical trials, in the treatment of acute stroke and head injuries

Also, the safety profile of citicoline is good, and there are no associated problems when the drug is used in this kind to patients

The aim of this study is to confirm the efficacy and safety of citicoline in patients with moderate-to-severe acute ischemic stroke in Egypt, according to the characteristics of the medical care in this country

DETAILED DESCRIPTION:
This is a Prospective Randomized Open-label trial with Blinded Evaluators, Citicoline will be administered in continuous Iv infusion in a dose of 2000 mg per day for the first week following AIS then by oral route for the next 5 weeks.

The number of patients needed for this proposal is 200 (100 per group): group 1 (citicoline): receiving citicoline and group 2 (control) not receiving citicoline. A 10% increase will be expected to avoid possible drop-outs.

Assessment scales:

Eligibility scale: NIHSS score ≥ 8. Outcome scales: modified Rankin Score (mRS) at 3 months Cutoff scores for mRS will be 0-2 as a cut-off point for a good outcome and 3-6 for a bad outcome.

Also, a record of all the side effects will be done. Any kind of adverse effect must be recorded by filling the CIOMS form.

Randomization: computer-generated randomization to either group.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders aged > 18 years.
* Patients must be treated within 24 hours of their initial stroke symptoms onset.
* Patients not eligible to receive rTPA.
* Patients with a measurable focal neurological deficit (NIHSS score ≥ 8) lasting for a minimum of 60 minutes. This deficit must persist from onset and up to the time of treatment without clinically significant improvement
* Patients must have a CT scan and/or conventional MRI compatible with the clinical diagnosis of acute ischemic stroke prior to being randomized.
* Patients must have an acute ischemic stroke with symptoms referrable to internal carotid territory.
* At inclusion, NIHSS score 8-15, with at least 2 of these points from sections 5 & 6 (motor).
* Immediately (i.e. minutes) pre-stroke, mRS ≤ 1. [History of past stroke does not, by itself, preclude study entrance].
* Women of childbearing potential must have a negative pregnancy test prior to enrolment.
* Signed informed consent (following a full explanation of the nature and purpose of this study, the patient or legal guardian(s) or representative(s) must consent to participate by signing the Informed Consent document

Exclusion Criteria:

* Patients eligible for rTPA treatment.
* Patients in coma: patients having a score of 2 or higher in the items regarding the level of consciousness in the NIHSS (1a).
* CT or conventional MRI evidence of any structural brain disorder other than ischemic stroke.
* History of ventricular dysrhythmias, acute myocardial infarction within 72 hours prior to enrolment, unstable angina, decompensated congestive heart failure or any other acute, severe, uncontrollable or sustained cardiovascular condition that, in the Investigator's opinion, may interfere with effective participation in the study.
* Previous disorders that may confound the interpretation of the neurological scales.
* Drug addiction-related disorders.
* Pre-existing dementia, when dementia implies a disability, measured as an score of 2 or higher in the previous mRS.
* Pre-existing medical condition that, in the Investigator's opinion, may interfere with the patient's suitability and participation in the study.
* Patients participating in another clinical trial or receiving a non-approved drug (clinical investigational drug) less than 30 days prior to screening.
* Patients under current treatment with citicoline.
* Prior (over past 3 months) or concomitant administration of other neuroprotectant drugs (such as nimodipine, vinponcetine, piracetam, cerebrolysin,…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with a good outcome using modified Rankin scale | 3 months
  the investigators will compare the percentage of patients with good outcomes in the citicoline group and control group according to the modified Rankin scale score.
  the modified Rankin scale (mRS) is a scale used to assess stroke outcomes, it ranges between 0 and 6 and the higher the score the worse the oucome.
  the investigators defined patients with good outcomes as patients with (mRS) at 3 months of (0-2), and patients with bad outcomes as those with mRS equals (3-6)

SECONDARY OUTCOMES:
Incidence of Citicoline-Emergent Adverse Events | 3 months
  the incidence of each adverse event related to citicoline will be calculated and recorded in CIOMS form and the investigators will compare the incidence of each side effect in the citicoline group and in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon appropriate request from authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon finishing study
Access Criteria: upon proper request from the author

REFERENCES:
- [Background] Adibhatla RM, Hatcher JF. Citicoline mechanisms and clinical efficacy in cerebral ischemia. J Neurosci Res. 2002 Oct 15;70(2):133-9. doi: 10.1002/jnr.10403. PMID 12271462
- [Background] Alvarez-Sabin J, Roman GC. The role of citicoline in neuroprotection and neurorepair in ischemic stroke. Brain Sci. 2013 Sep 23;3(3):1395-414. doi: 10.3390/brainsci3031395. PMID 24961534
- [Background] Cho HJ, Kim YJ. Efficacy and safety of oral citicoline in acute ischemic stroke: drug surveillance study in 4,191 cases. Methods Find Exp Clin Pharmacol. 2009 Apr;31(3):171-6. doi: 10.1358/mf.2009.31.3.1364241. PMID 19536360
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/12271462
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/24961534
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/19536360